CLINICAL TRIAL: NCT05527886
Title: Acute Effects of Dynamic Stretching, Plyometrics, and Loading on Achilles Tendon Properties and Performance Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Dakota (Other)
Responsible Party: Principal Investigator, Matt Dewald, Assistant Professor, University of South Dakota
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 22-211
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Tendon Injuries
MeSH Terms: conditions — Tendon Injuries | interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The researchers collecting data will be blinded to the intervention provided
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Randomized AAROM, Slow Load, or Plyometric intervention
  Interventions: Other: AAROM; Other: Slow Load; Other: Plyometric
- Group 2 (Experimental): Randomized AAROM, Slow Load, or Plyometric intervention
  Interventions: Other: AAROM; Other: Slow Load; Other: Plyometric
- Group 3 (Experimental): Randomized AAROM, Slow Load, or Plyometric intervention
  Interventions: Other: AAROM; Other: Slow Load; Other: Plyometric

INTERVENTIONS:
Other: AAROM — AAROM with knee to wall exercise, 3x30 reps
Other: Slow Load — Single leg heel raise, 3x10 reps
Other: Plyometric — Double leg 5 inch wall hops, 3x10 sec

SUMMARY:
The study will be looking at acute changes in Achilles tendon properties and changes in a vertical single leg hop following an exercise intervention. The three exercise interventions will be randomized and take place on separate days 1 week apart. The three exercise interventions are AAROM, slow load, and plyometrics.

DETAILED DESCRIPTION:
The purpose of the study is to determine if there are acute changes in Achilles tendon properties and changes in performance based on what tendon exercise intervention is being used. About 70 people will take part in this research.

ELIGIBILITY:
Inclusion Criteria:

* College student

Exclusion Criteria:

* Unable to complete interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Achilles Tendon Stiffness | immediately
  A myotonometer will measure the stiffness in N/m.
Achilles Tendon Natural Oscillation | immediately
  A myotonometer will measure the natural oscillation frequency in Hz.
Achilles Tendon Logarithmic Decrement | immediately
  A myotonometer will measure logarithmic decrement, which is a measure of elasticity.
Achilles Tendon Mechanical Stress Relaxation Time | immediately
  A myotonometer will measure mechanical stress relaxation time in ms.
Achilles Tendon Creep | immediately
  A myotonometer will measure creep in De.

SECONDARY OUTCOMES:
Single-leg drop jump vertical | immediately
  Single-leg vertical drop jump from 4-inch box with knee locked in extension will be measured in cm. A higher jump is considered better.
Reactive Strength Index | immediately
  Reactive Strength Index will be measured as an AU, the higher the better.
Flight Time | immediately
  Flight time will be measured in ms, the higher the better.
Contact Time | immediately
  Contact time will be measured in ms, the lower the better.
Limb Stiffness | immediately
  Limb stiffness will be measured in kN/m, generally the higher the better.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanford Coyote Sport Center, Vermillion, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: If required with the publication, a link to de-identified data will be provided.
Access Criteria: IPD will be available upon request